CLINICAL TRIAL: NCT06331299
Title: A Phase 3, Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of UGN-103, a Novel Formulation of UGN-102, for the Treatment of Patients With Low-grade (LG) Non-muscle Invasive Bladder Cancer (NMIBC) at Intermediate-risk (IR) of Recurrence
Brief Title: A Phase 3 Study of UGN-103 for Treatment of Patients With Low-grade Intermediate-risk Non-muscle Invasive Bladder Cancer
Acronym: UTOPIA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL013
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Urothelial Carcinoma Bladder
Keywords: Non-muscle invasive bladder cancer; Low-grade non-muscle invasive bladder cancer; Intermediate-risk non-muscle invasive bladder cancer; NMIBC; UGN-103; UGN-102; Mitomycin
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UGN-103 (Experimental): Patients will receive UGN-103 (75 mg mitomycin) once weekly for 6 weeks (a total of 6 doses).
  Interventions: Drug: UGN-103

INTERVENTIONS:
Drug: UGN-103 — UGN-103 consists of mitomycin and sterile hydrogel (a proprietary thermally responsive gel) that is used to reconstitute mitomycin before instillation. The reverse thermal properties of UGN-103 allow for local administration of mitomycin as a liquid under chilled conditions, with subsequent conversion to a semi-solid gel depot following instillation into the bladder.
  Other Names: UGN-103 (mitomycin) for intravesical solution

SUMMARY:
This Phase 3, single-arm, multicenter study will evaluate the efficacy and safety of UGN-103, a novel formulation of UGN-102, instilled in the urinary bladder of patients with low-grade non-muscle invasive bladder cancer (LG-NMIBC).

DETAILED DESCRIPTION:
Eligible patients will be treated with UGN-103 once weekly for 6 weeks (a total of 6 doses).

Efficacy will be assessed by the complete response rate (CRR) at the 3-month Visit (approximately 3 months after the first instillation). Response will be determined based on visual observation (white light cystoscopy), histopathology of any remaining or new lesions by central pathology lab (if applicable), and interpretation of urine cytology by central pathology lab.

Patients who have a complete response (CR) at the 3-month Visit, defined as having no detectable disease (NDD) in the bladder, will enter the Follow-up Period of the study. During the Follow-up Period, patients will return to the clinic every 3 months for evaluation of response. Patients will remain on study until disease recurrence, disease progression, death, or the last patient completes 12 months of follow-up (ie, 12 months after the 3-month Visit), whichever occurs first.

Patients who have a non-complete response (NCR) at the 3-month Visit will undergo investigator designated standard of care (SOC) and have a separate End of Study (EOS) Visit performed.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and the protocol.
2. Patient who has LG-NMIBC (Ta) histologically confirmed by cold cup biopsy at Screening or within 8 weeks before Screening.
3. History of at least 1 prior episode of NMIBC. Note: This refers to a previous episode(s) and not to the current episode for which the patient is being screened.
4. Has intermediate-risk disease, defined as having 1 or 2 of the following:

   * Presence of multiple tumors.
   * Solitary tumor > 3 cm.
   * Early or frequent recurrence (≥ 1 occurrence of LG-NMIBC within 1 year of the current diagnosis at the initial Screening Visit).
5. Negative voiding cytology for high-grade (HG) disease within 8 weeks before Screening.
6. Has adequate organ and bone marrow function as determined by routine laboratory tests:

   * Leukocytes ≥ 3,000/μL.
   * Absolute neutrophil count ≥ 1,500/μL.
   * Platelets ≥ 100,000/μL.
   * Hemoglobin ≥ 9.0 g/dL.
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN).
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN.
   * Alkaline phosphatase (ALP) ≤ 2.5 × ULN.
   * Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min.
7. Has an anticipated life expectancy of at least the duration of the trial.
8. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Women of childbearing potential (defined as premenopausal women who have not been sterilized), including female patients and female partners of male patients, must be willing to use 2 acceptable forms of effective contraception from enrollment through 6 months post-treatment.

Exclusion Criteria:

1. Received Bacillus Calmette-Guérin (BCG) treatment for urothelial carcinoma (UC) within the previous 1 year.
2. History of HG bladder cancer (papillary or carcinoma in situ) in the past 2 years.
3. Known allergy or sensitivity to any component of the study treatment (including excipients) that in the investigator's opinion cannot be readily managed.
4. Clinically significant urethral stricture that would preclude passage of a urethral catheter.
5. History of:

   * Neurogenic bladder.
   * Active urinary retention.
   * Any other condition that would prohibit normal voiding.
6. Past or current muscle invasive bladder cancer (ie, T2, T3, T4) or metastatic UC.
7. Current tumor stage of T1.
8. Concurrent upper tract urothelial carcinoma (UTUC).
9. Evidence of active urinary tract infection (UTI) that in the investigator's opinion cannot be treated and resolved prior to biopsy and/or administration of study treatment.
10. Is pregnant or breastfeeding.
11. Has an underlying substance abuse or psychiatric disorder such that, in the opinion of the investigator, the patient would be unable to comply with the protocol.
12. History of prior treatment with an intravesical chemotherapeutic agent in the past 2 years except for a single dose of chemotherapy immediately after any previous transurethral resection of bladder tumors (TURBT).
13. Has participated in a study with an investigational agent or device within 30 days of enrollment.
14. Has previously participated in a study in which they received UGN-102.
15. Has any other active malignancy requiring treatment with systemic anticancer therapy (eg, chemotherapy, immunotherapy, radiation therapy). Superficial cancers such as cutaneous basal cell or squamous cell carcinomas that can be treated locally are allowed.
16. Has any other clinically significant medical or surgical condition that in the investigator's opinion could compromise patient safety or the interpretation of study results.
17. Where applicable per country regulation, the patient must not be currently committed to an institution by virtue of an order issued by either judicial or administrative authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | 3 months
  CRR is defined as the proportion of patients who achieved CR at the 3-month Visit.

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 21 months
  DOR is defined as the time from the date of evidence of CR at the 3-month Visit to the earliest date of recurrence or progression or death due to any cause, whichever occurred first.
Durable complete response (DCR) rate | Up to 21 months
  DCR rate at scheduled disease assessment time points, defined as the proportion of patients who achieved CR at the 3-month Visit and maintained CR (ie, no detectable disease) up to that particular follow-up disease assessment.
Incidence of treatment-emergent adverse events (TEAEs), serious TEAEs, TEAEs of special interest, and abnormal clinical laboratory test results (hematology and serum chemistry) | Up to 21 months
  The number of patients with each type of event will be summarized.
Mitomycin plasma concentrations | 0 (pre-instillation), 0.5, 1, 2, 3, 4, 5, and 6 hours after the first instillation of UGN-103.
  Mitomycin plasma concentrations will be assessed in a subset of patients treated with UGN-103
Mitomycin maximum plasma concentration (Cmax) | 0 (pre-instillation), 0.5, 1, 2, 3, 4, 5, and 6 hours after the first instillation of UGN-103.
  Mitomycin Cmax will be assessed in a subset of patients treated with UGN-103

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mirkin, MD, Study Director — UroGen Pharma
Locations (48):
- United States (17):
  - Loma Linda University Medical Center, Loma Linda, California
  - Genesis Research, LLC, San Diego, California
  - The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Peachtree Clinical Solutions, Powder Springs, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Minnesota Urology - Metro Urology - Woodbury, Woodbury, Minnesota
  - Garden State Urology, Morristown, New Jersey
  - Great Lakes Physician dba WNYU, Cheektowaga, New York
  - AccuMed Research Associates, Garden City, New York
  - Crystal Run Healthcare, Middletown, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, New York, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates P.C. - Nashville, Nashville, Tennessee
  - Houston Metro Urology (HMU) - Southwest Location, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Spokane Urology, P.S., Spokane, Washington
- Bulgaria (7):
  - Multiprofile Hospital for Active Treatment "Dr. Tota Venkova", Gabrovo, Department of Urology, Gabrovo, Gabrovo
  - University Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski", Pleven, Urology Clinic, Pleven, Pleven Province
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv, Clinic of Urology, Plovdiv, Plovdiv Province
  - University Multiprofile Hospital for Active Treatment, Plovdiv, Clinic of Urology, Plovdiv, Plovdiv Province
  - University Multiprofile Hospital for Active Treatment 'Kanev', Ruse, Department of Urology, Rousse, Ruse Province
  - Multiprofile Hospital for Active Treatment - Shumen, Department of Urology, Shumen, Shumen Province
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I. Pirogov", Sofia, Urology Clinic, Sofia, Sofia-Grad
- Estonia (4):
  - West Tallinn Central Hospital Ltd., Department of Urology, Tallinn, Harju
  - North Estonia Medical Centre Foundation Ltd., Tallinn, Harju
  - East Viru Central Hospital, Surgery Clinic, Kohtla-Järve, Ida-Virumaa
  - Tartu University Hospital, Surgery Clinic, Department of Urology and Kidney Transplantation, Tartu, Tartu County
- Georgia (5):
  - LLC "Todua Clinic", Tbilisi
  - Geo Hospitals LLC, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic LLC, Tbilisi
  - LTD MMT Hospital, Tbilisi
  - JSC Jerarsi, Tbilisi
- Latvia (4):
  - Daugavpils Regional Hospital, Urology Department, Daugavpils
  - Liepajas Regional Hospital, Urology Department, Liepāja
  - P. Stradins Clinical University Hospital, Center for Urology, Riga
  - LLC Riga East University Hospital, Clinic of Urology and Oncologic Urology, Riga
- Romania (6):
  - Bihor County Emergency Clinical Hospital, Oradea, Bihor County
  - Brasov County Emergency Clinical Hospital, Department of Urology, Brasov, Brașov County
  - Craiova County Emergency Clinical Hospital, Department of Urology, Craiova, Dolj
  - SC Clinica Polisano Hospital, Sibiu, Sibiu County
  - Colentina Clinical Hospital, Department of Urology, Bucharest
  - "Prof. Dr. Th. Burghele" Clinical Hospital, Department of Urology III, Bucharest
- Spain (5):
  - University Hospital Virgen de la Victoria, Málaga, Andalusia
  - Puigvert Foundation, Barcelona, Catalonia
  - University Hospital Foundation Jimenez Diaz, Madrid, Madrid
  - University Hospital 12 de Octubre, Madrid, Madrid
  - La Paz University Hospital, Madrid, Madrid